CLINICAL TRIAL: NCT01362114
Title: Phase 4 Study of The Effect of Sihogayonggolmoryeo-tang on the Anxiety of Hwa-byung : A Randomized, Double Blind, Placebo-control Trial
Brief Title: The Effect of Sihogayonggolmoryeo-tang on the Anxiety of Hwa-byung
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, In-Chul Jung, Professor of Oriental Hospital of Daejon University, Korea Health Industry Development Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B080009
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Hwa-byung
Keywords: Hwa-byung; Sihogayonggolmoryeo-tang; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sihogayonggolmoryeo-tang extract (Experimental): * name of product: 'SIHOGAYONGGOLMORYU TANG EXTRACT GRAN'
  * standard code for item: 200005676
  * shape, type: extract(brown)
  * usage, content: adults;three times a day, each taken before or between meals
  * dose, standard: 2.5g for each sack, capsulated
  * storage : airtight container, stored in room temperature
  * expiration date : 36months after manufacture
  * macufacturing company: KyungBangnShinYak inc.
  Interventions: Drug: SIHOGAYONGGOLMORYU TANG EXTRACT GRAN
- Placebo; corn flour, (Placebo Comparator): * raw material: total contents(500㎎); cornstarch 50.0%(250.0㎎), 당수화물 49.45%(247.25㎎), caramel pigment 0.5%(2.5㎎), SsangHwa fragrance 0.05%(0.25㎎)
  * shape, type: extract(brown)
  * usage, dose: adults: three times a day, 1 sack before or between meals
  * dose, standard: 2.5g for each sack, capsulated
  * storage : airtight container, stored in room temperature
  * expiration date : 36 months after manufacture
  * manufacturing company: KyungBangnShinYak inc.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SIHOGAYONGGOLMORYU TANG EXTRACT GRAN — three times a day, AC 30 min., 4 capsules taken each time (4capsules=2.5g), 8 weeks
  Other Names: standard code for item: 200005676
  Arms: Sihogayonggolmoryeo-tang extract
Other: Placebo — three times a day, AC 30 min., 4 capsules taken each time (4capsules=2.5g), 8 weeks.
  Arms: Placebo; corn flour,

SUMMARY:
In this randomized, double blinded, Placebo-control Trial, the investigators planned to give Sihogayonggolmoryeo-tang extract or controlled medication on the Anxiety of Hwa-byung.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 20-65
* subjects who meet structured interview criteria for Hwa-Byung Diagnosis
* subjects who have axiety (more than 17 score in HAMA)

Exclusion Criteria:

* duration of illness less than 6 months
* current or past history of delusions, hallucination
* past history of at least one manic episode, hypomanic episode, or mixed episode
* current or past history of alcohol abuse or alcohol dependence history
* taking substances(e.g. steroids) which might affect symptoms
* medical conditions(e.g. hyperthyroidism, hypothyroidism, heart disease) that might affect symptoms
* current with hepatoma, hepatic cirrhosis, chronic renal failure, congestive heart failure
* pregnancy, lactation, women not using medically accepted means of birth control
* considered not apt to carry out clinical trial

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-05 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale(HAM-A) | 8 weeks
  The HAM-A (Hamilton Anxiety Scale) is a widely used interview scale that measures the severity of a patient's anxiety, based on 14 parameters, including anxious mood, tension, fears, insomnia, somatic complaints and behavior at the interview.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory(STAI) | 8 weeks
  The State-Trait Anxiety Inventory (STAI) was initially conceptualized as a research instrument for the study of anxiety in adults. It is a self-report assessment device which includes separate measures of state and trait anxiety.
Beck Depression Inventory(BDI) | 8 weeks
  BDI is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression. Each question has a set of at least four possible answer choices, ranging in intensity. When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity.
WHO Quality of Life Abbreviated(WHOQOL-BREF) | 8 weeks
  Quality of life is used to evaluate the general well-being of individuals and societies.
Heart Rate Variability(HRV) | 8 weeks
  Heart rate variability (HRV) is a physiological phenomenon where the time interval between heart beats varies. It is measured by the variation in the beat-to-beat interval.
likert scale | 8 weeks
  This scale is used to evaluate the degree of Hwa-byung's major symptom by 5 point measure. (0,1,2,3,4)
Hwa-byung scale | 8 weeks
  This scale is used for self report to evaluate the Hwa-byung's emotional symptoms, physical symptoms and personality traits by 5 point.(0,1,2,3,4).
State-Trait Anger Expression Inventory (STAXI) | 8 weeks
  The State-Trait Anger Expression Inventory is a inventory which measures the intensity of anger as an emotional state (State Anger) and the disposition to experience angry feelings as a personality trait (Trait Anger). Items consist of 4-point scales that assess intensity of anger at a particular moment and the frequency of anger experience, expression, and control.
Insomnia Severity Index (ISI) | 8 weeks
  The Insomnia Severity Index is a series of questions, seven in total, designed by medical professionals to help gauge the seriousness of a person's insomnia. The seven questions have numerical value, and the total is added up at the end of the process to give a total that symbolizes the seriousness of the problem
Instrument of Oriental Medical Evaluation for Hwa-Byung | 8 weeks
  Instrument of Oriental Medical Evaluation for Hwa-Byung is a standard scale to evaluate for Oriental Medical cure in Hwa-Byung

CONTACTS AND LOCATIONS:
Overall Officials: In-Chul Jung, Ph.D, Principal Investigator — Oriental Hospital of Daejon University
Locations (1):
- Oriental Hospital of Daejon University, Daejeon, Choong-Chung-Do, South Korea